CLINICAL TRIAL: NCT00864487
Title: A Study to Examine the Potential Effect of Rifampin on the Pharmacokinetics of Neratinib When Administered Concomitantly to Healthy Subjects
Brief Title: Study Evaluating The Potential Effect Of Rifampin On The Pharmacokinetics Of Neratinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3144A1-1110
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Neratinib alone
  Interventions: Drug: Neratinib
- 2 (Experimental): Neratinib plus rifampin
  Interventions: Drug: Neratinib

INTERVENTIONS:
Drug: Neratinib — HKI-272

SUMMARY:
The purpose of this study is to examine whether co-administration of rifampin with neratinib has an effect on the pharmacokinetics (how the body absorbs, distributes, metabolizes and/or excretes) of neratinib.

ELIGIBILITY:
Inclusion criteria:

* Healthy men or women (of non childbearing potential)
* Ages 18 to 50 years old.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (plasma blood concentrations) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (1):
- Miami, Florida, United States